CLINICAL TRIAL: NCT05922878
Title: A Randomized, Double-Blind, Placebo-Controlled Study of ALTO-300 With an Open-Label Extension in Adults With Major Depressive Disorder
Brief Title: Study of ALTO-300 in MDD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Alto Neuroscience (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALTO-300-201
Record Dates: First submitted 2023-05-26; First posted 2023-06-28 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-06

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- ALTO-300 (Experimental): Participants will receive ALTO-300 capsule once daily in the evening, from Day 1 to Day 42 in double blind (DB) treatment period. Eligible participants who will enter the open-label (OL) treatment period will receive ALTO-300 capsule once daily in the evening from OL baseline until the end of OL period/early termination visit (Up to 8 weeks).
  Interventions: Drug: ALTO-300
- Placebo (Placebo Comparator): Participants will receive matching placebo capsule once daily in the evening, from Day 1 to Day 42 in double blind (DB) treatment period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ALTO-300 — ALTO-300 capsule QD
  Arms: ALTO-300
Drug: Placebo — Placebo capsule QD
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine efficacy differences between ALTO-300 and placebo, used adjunctively to an antidepressant, related to patient characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of moderate to severe major depressive disorder (MDD)
* At Visit 1, currently taking a single SSRI, SNRI, or bupropion for at least 6 weeks with no dose modifications in the past 2 weeks by Visit 2
* Willing to comply with all study assessments and procedures
* Must not be pregnant or breastfeeding at time of enrollment or throughout study

Exclusion Criteria:

* Evidence of unstable medical condition
* Nightly use of sleep medication
* Diagnosed bipolar disorder, psychotic disorder, or dementia
* Current moderate or severe substance use disorder
* Has a history of hypersensitivity or allergic reaction to ALTO-300 or any of its components/excipients
* Concurrent or recent participation in another clinical trial for mental illness involving an investigational product or device

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 321 (Estimated)
Dates: Start 2023-06-08 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
To assess efficacy of adjunctive ALTO-300 versus placebo on symptoms of MDD in a pre-defined subgroup of participants as measured by the change over time up to week 6 in the Montgomery-Åsberg Depression Rating Scale (MADRS). | Change over time for up to week 6
  MADRS is a clinician-administered scale designed to measure depression severity and detects changes due to antidepressant treatment. The MADRS evaluates the following 10 items: apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts. Each item is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total possible score of 60. Higher scores represent a more severe condition.

SECONDARY OUTCOMES:
To assess efficacy of adjunctive ALTO-300 versus placebo on symptoms of MDD in all randomized participants as measured by the change over time up to week 6 in the Montgomery-Åsberg Depression Rating Scale (MADRS) | Change over time for up to week 6
  MADRS is a clinician-administered scale designed to measure depression severity and detects changes due to antidepressant treatment. The MADRS evaluates the following 10 items: apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts. Each item is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total possible score of 60. Higher scores represent a more severe condition.
To assess efficacy of adjunctive ALTO-300 versus placebo for MDD as measured by the change over time up to week 6 in response (>50% improvement from baseline) rates based on the MADRS | Change over time for up to week 6
  MADRS is a clinician-administered scale designed to measure depression severity and detects changes due to antidepressant treatment. The MADRS evaluates the following 10 items: apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts. Each item is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total possible score of 60. Higher scores represent a more severe condition.
To evaluate the safety of ALTO-300 during both the OL and DB periods of the study as measured by the assessment of the incidence, severity, and relatedness of Adverse Events. | Assessed from Day 1 to Week 14
  Incidence, severity, and relatedness of Adverse Events
To evaluate the safety of ALTO-300 during both the OL and DB periods of the study as measured by the assessment of Heart Rate. | Assessed from Day 1 to Week 14
  Assessment of Heart Rate
To evaluate the safety of ALTO-300 during both the OL and DB periods of the study as measured by the assessment of Weight. | Assessed from Day 1 to Week 14
  Assessment of Weight
To evaluate the safety of ALTO-300 during both the OL and DB periods of the study as measured by the assessment of Blood Pressure. | Assessed from Day 1 to Week 14
  Assessment of Blood Pressure
To evaluate the safety of ALTO-300 during both the OL and DB periods of the study as measured by the assessment of suicidality with the Concise Health Risk Tracking Self-Report,12 item scale (CHRT-SR12). | Assessed from Day 1 to Week 15
  The CHRT is a brief, self-report measure that systematically assesses both suicidal thinking and associated thoughts that may indicate the propensity for suicidal acts. The CHRT-SR12 is a 12 item scale. The patient assigns a score of 0-4 for each item of the scale, allowing for a total score of 0 to 48, with the higher score signifying more severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Savitz, MD, PhD, Study Director — Alto Neuroscience
Locations (45):
- United States (45):
  - Site 200, Phoenix, Arizona
  - Site 189, Phoenix, Arizona
  - Site 187, Yuma, Arizona
  - Site 193, Rogers, Arkansas
  - Site 218, Bellflower, California
  - Site 217, Glendale, California
  - Site 335, Lafayette, California
  - Site 209, Los Angeles, California
  - Site 219, Mather, California
  - Site 194, Mission Viejo, California
  - Site 197, Temecula, California
  - Site 203, Colorado Springs, Colorado
  - Site 349, Evergreen, Colorado
  - Site 214, Norwalk, Connecticut
  - Site 159, Clermont, Florida
  - Site 225, Miami Gardens, Florida
  - Site 190, Miami Lakes, Florida
  - Site 161, Okeechobee, Florida
  - Site 221, Tampa, Florida
  - Site 220, West Palm Beach, Florida
  - Site 224, Savannah, Georgia
  - Site 208, Snellville, Georgia
  - Site 119, Boise, Idaho
  - Site 310, Chicago, Illinois
  - Site 201, Marrero, Louisiana
  - Site 198, Monroe, Louisiana
  - Site 215, Jackson, Mississippi
  - Site 344, Las Vegas, Nevada
  - Site 114, Albuquerque, New Mexico
  - Site 191, Rochester, New York
  - Site 192, Staten Island, New York
  - Site 199, Hickory, North Carolina
  - Site 202, Cincinnati, Ohio
  - Site 195, Oklahoma City, Oklahoma
  - Site 216, Allentown, Pennsylvania
  - Site 350, Media, Pennsylvania
  - Site 352, Moosic, Pennsylvania
  - Site 102, Dallas, Texas
  - Site 347, Fort Worth, Texas
  - Site 148, Fort Worth, Texas
  - Site 206, Missouri City, Texas
  - Site 353, Plano, Texas
  - Site 196, Richmond, Texas
  - Site 207, Clinton, Utah
  - Site 211, Roanoke, Virginia